CLINICAL TRIAL: NCT06582433
Title: The Effectiveness of Solution-Focused Counseling in Managing Menopausal Symptoms
Brief Title: Solution-focused Counseling for Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-77192459-050.99-338559
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Menopause; Menopause Related Conditions; Menopausal Depression
Keywords: Menopause; Menopausal Symptoms; Solution-focused counseling
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- İntervention group (Experimental): Pre-Procedure: Women who meet the inclusion criteria will be divided into experimental and control groups using simple randomization method. Before the procedure, both groups will fill out the Personal Information Form (PIF), Psychological Well-being Scale (PWS), Menopausal Symptoms Assessment Scale (MSAS), and Menopause Attitude Assessment Scale(MASS) (1st Measurement).
  During the Procedure: Women in the experimental group will receive Solution-Focused Counseling (SFC) by the researcher. SFC will be conducted individually once a week, in a total of 6 sessions, with each session lasting 60 minutes.
  Post-Procedure: One week after the completion of SFC sessions, both groups will fill out PWS, MSAS, and MAAS again (2nd Measurement).
  Follow-Up Two Months Later: Two months later, both groups will fill out PWS, MSAS, and MAAS again to evaluate whether the effects of SFC are still present (Follow-Up Measurement).
  Interventions: Other: Intervention
- Control group (No Intervention): Before the procedure, women will be asked to fill out a Personal Information Form (PIF), Psychological Well-being Scale (PWS), Menopause Symptoms Assessment Scale (MSAS), and Menopause Attitude Assessment Scale (MAAS) (1st Measurement). Women in the control group will be provided with information about routine menopausal symptoms. 2 months later, the 2nd Measurement will be taken. After the follow-up measurement is taken for the control group, counseling will be provided to women according to their needs (addressing problems, answering questions, providing information as needed).

INTERVENTIONS:
Other: Intervention — 1. Process: implementation of pre-tests
  2. Process: Solution-focused counseling, 60 minutes once a week for a total of 6 sessions
  3. Final test after 2 months
  Other Names: Experimental Group
  Arms: İntervention group

SUMMARY:
This research will be conducted in a prospective pre-test post-test measurement randomized controlled experimental design. The population of the study consists of women who have entered menopause and live in Karabük. The research sample size was calculated considering the literature information that in experimental studies each group should consist of at least 30 individuals, taking into account the power of the test with G*Power 3.1 Program. It was calculated that at least 32 observations are needed in both the experimental and control groups to reach a power level of 90% at a significance level of 5% with an effect size of 0.75, and the sample size of the study was calculated as 64 women. The data of the study will be collected using the "Personal Information Form", "Psychological Well-being Scale", "Menopausal Symptoms Evaluation Scale" and "Menopause Attitude Evaluation Scale".

WORKFLOW

Pre-procedure:

* Women who meet the inclusion criteria for the study will be divided into experimental and control groups using simple randomization method.
* Before the procedure, women in both groups will fill out the PIF, PWBS, MSES, and MAES (1st Measurement).

During the procedure:

At this stage, Solution-Focused Counseling (SFC) will be used on women in the experimental group by the researcher. SFC sessions for patients will be held individually, once a week, with a total of 6 sessions that may have deviations of 2-3 days before or after the previous session. Each session is planned to last 60 minutes. Counseling for patients will be conducted in a comfortable environment. At this stage, women in the control group will be given information on typical menopausal symptoms.

Post-procedure:

One week after the completion of SFC sessions, the PIF, PWBS, MSES, and MAES will be filled out by the experimental and control groups (2nd Measurement).

Follow-up evaluation after 2 months:

Two months after the completion of SFC sessions, the PIF, PWBS, MSES, and MAES will be applied to the experimental and control groups (Follow-up Measurement) to determine whether the results of the applied SFC are continuing.After monitoring measurements are taken on the control group, counseling will be provided to women according to their needs (addressing issues, answering questions, informing them according to their needs).

DETAILED DESCRIPTION:
The aim of this research is to examine the effectiveness of solution-focused counseling in managing menopausal symptoms and to investigate the impact of this approach on the attitudes and psychological well-being of women in the menopausal period.

H1: Solution-focused counseling affects the evaluation of menopausal symptoms in women in the menopausal period.

H2: Solution-focused counseling leads to changes in attitudes towards menopause in women in the menopausal period.

H3: Solution-focused counseling affects the level of psychological well-being of women in the menopausal period.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study
* Being a woman
* Having been diagnosed with menopause for at least 1 year

Exclusion Criteria:

* Leaving work halfway through without filling out surveys or scales even though you stayed to work
* Having any barriers to communication
* Having received a psychiatric diagnosis

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — period of menopause
Enrollment: 44 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
prevention | One session per week, each session is 90 minutes, a total of 6 sessions.
  Menopausal complaints

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Karabük Province, Turkey (Türkiye)